CLINICAL TRIAL: NCT05665400
Title: A Cross-sectional, Interventional, Exploratory Clinical Study for the Development of a Device (Lovelace) for Antepartum Fetal Monitoring
Brief Title: A Clinical Study for the Development of a Device (Lovelace) for Antepartum Fetal Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloom Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LOV-01-2022-EU
Record Dates: First submitted 2022-06-21; First posted 2022-12-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Fetal Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bloomlife Lovelace FT (Experimental)
  Interventions: Device: Bloomlife Lovelace FT

INTERVENTIONS:
Device: Bloomlife Lovelace FT — Bloomlife Lovelace FT is a non-invasive, wireless, external measurement system used to measure accelerometer and electrophysiological signals on pregnant women with a singleton pregnancy, by acquiring biopotential signals from abdominal surface electrodes.

SUMMARY:
Bloomlife Lovelace FT is a non-invasive, wireless, external measurement system used to measure accelerometer and electrophysiological signals on pregnant women with a singleton pregnancy, by acquiring biopotential signals from abdominal surface electrodes.

In this study, Bloomlife Lovelace FT is used to collect the dataset needed for the development of a future product (Bloomlife Lovelace) for the monitoring of fetal heart rate, maternal heart rate and uterine activity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman ≥ 18 years old
* Gestational age greater or equal to 24 weeks and 0 days
* Singleton pregnancy
* Ability to read and understand Dutch
* Willingness to participate in the study

Exclusion Criteria:

* Implanted pacemaker or any other implanted electrical device
* History of allergies to skin adhesives
* Irritated or lesioned skin at the Bloomlife Lovelace FT electrodes locations
* Contraindication to the use of CTG based on physician's decision (e.g. due to preterm contractions)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Extent of agreement between Bloomlife Lovelace FT and CTG in fetal heart rate | 1 hour
  Bland-Altman analysis, based on a 95% limits of agreement.
Extent of agreement between Bloomlife Lovelace FT and CTG in maternal heart rate | 1 hour
  Bland-Altman analysis, based on a 95% limits of agreement.
Performance metrics of Contraction Detection with Bloomlife Lovelace FT | 1 hour
  Sensitivity, False Event Rate, Positive Percentage Agreement, Negative Percentage Agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Van Holsbeke, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided